CLINICAL TRIAL: NCT06824558
Title: Effect of Virgin Mary Herb Used in Birth on Duration, Pain and Fear of Childbirth: A Randomized Controlled Trial
Brief Title: The Effects of the Use of Virgin Mary Herb in Childbirth
Acronym: EVMHUBDPFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Tuğba YILMAZ ESENCAN, assistant professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Virgin Mary Herb Used in Birth
Record Dates: First submitted 2025-01-23; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Pain During Labour; Fear of Childbirth
Keywords: Anastatica Hierochuntica

STUDY DESIGN:
Intervention Model Description: The researcher will provide the Virgin Mary herb. A Virgin Mary herb plant will be used for each pregnant woman. The herb will be weighed with a precision scale to ensure that it is the same size and weight. The intervention group will be asked to fill out the same data collection tools by watching 100 grams of Virgin Mary herb in a standard wide-mouthed glass bowl at 50 degrees and put in a container full of water. The monitoring period of the Virgin Mary herb will be recorded in the Virgin Mary Herb Monitoring Form and the visuals during this time will be photographed and monitored through this form. At the same time, the labor will be monitored with the midwifery care provided by the researcher midwife throughout the progress of the labor. The pregnant woman will be told to imagine that her cervix is opening in this way while watching the herb opening. The details regarding the application (monitoring period of Anastatica Hierochuntica) will be recorded by
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- primiparous pregnant (Sham Comparator): Control group: Normal midwifery care is applied during birth and no other care is applied. Pregnant women are not shown the blossoming of the Virgin Mary plant in water as in the intervention group.
  Interventions: Other: primiparous pregnant
- primiparous pregnant woman following virgin mary (Active Comparator): Pregnant women in the intervention group were shown the herb Mary taken in water during birth and also received midwifery care.
  Interventions: Other: primiparous pregnant woman following virgin mary

INTERVENTIONS:
Other: primiparous pregnant woman following virgin mary — It is thought that the application of the motherwort during birth shortens the duration of labor and reduces pain and fear during birth. In the study, the pregnant women in the intervention group watched the opening of the motherwort in water during birth.
  Arms: primiparous pregnant woman following virgin mary
Other: primiparous pregnant — Only midwifery care was applied to pregnant women in the control group.
  Arms: primiparous pregnant

SUMMARY:
This is a study to see if the use of virgin mary herb during birth has an effect on fear, pain and duration during birth. Virgin mary herb is a dry plant and it is believed that when added to water during birth, it makes birth easier.

DETAILED DESCRIPTION:
Objective: Midwives mostly develop nonpharmacological methods to cope with fear and pain management during birth in order not to interfere with the flow of birth. There are limited studies on traditional birth methods in Turkey. The aim of this study is to examine the effect of the use of the Virgin Mary Herb, one of the traditional methods applied during birth, on fear of birth and pain felt during birth. Material and Method: The universe of the study consists of all pregnant women who were admitted to the Birth Unit of a City Hospital in Istanbul between March 2023 and December 2023. A power analysis was conducted to determine the number of people to be included in the study sample. The power of the test was calculated with the G*Power 3.1 program. In order to exceed the 95% value in determining the power of the study; a total of 84 people, 42 people in groups, should be reached at a significance level of 5% and an effect size of 0.732 (df=82; t=1.66). The study aimed to reach a total of 100 people, with the condition of including 50 people in each group, considering the high power of the test and the losses. Data were collected between September 5, 2024 and December 31, 2024. 50 intervention groups and 50 control groups were included in the study, and all pregnant women received midwifery care. The intervention group was additionally shown the opening of the Virgin Mary Herb in water.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Being able to understand and speak Turkish,
* Being primiparous,
* Not having a chronic disease,
* Having completed the 37th week of pregnancy,
* Not having passed the 42nd week of pregnancy,
* Being in a cephalic presentation,
* Having reached 4cm cervical dilatation,

Exclusion Criteria:

* Multiparous pregnancy,
* Application of labor induction,
* Being a high-risk pregnancy,
* Having received childbirth preparation training,
* Being an immigrant,
* Use of non-pharmacological methods other than Virgin Mary

Ages: 18 Days to 45 Days | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — The study was conducted on primiparous pregnant women.
Enrollment: 100 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Fear Scale | After the pregnant woman started labor(when cervical dilatation was 4cm and above), the application was started. Labor lasted on average 24 hours.During this time the pregnant woman was assessed 3 times
  It is a scale developed by Serçekuş, İşbir and İnci in 2017. The Turkish form of the Fear of Childbirth Scale is a measurement tool that can accurately measure fear during childbirth, can be applied to Turkish culture, and is suitable in terms of language and content validity. The scale is a practical and fast tool to determine the degree of fear during childbirth and has been recommended to be used to determine the degree of fear of women in delivery rooms. Detection of fear during childbirth can allow continuous supportive care (emotional, informative support, relaxation, etc.) during childbirth, allowing the woman to have a better birth experience. Therefore, the Fear of Childbirth Scale can be used by professionals to determine the degree of fear of women in delivery rooms. The scale consists of 10 questions. Each question was scored between 1 and 10. The higher the score, the higher the fear.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | After the pregnant woman started labor(when cervical dilatation was 4cm and above), the application was started.Labor lasted on average 24 hours.During this time the pregnant woman was assessed 3times
  VAS was developed to be used in converting some values that cannot be measured quantitatively into numerical values. In VAS, where pain intensity is evaluated, pain intensity is graded between 0 and 10 points. "No pain" is graded as 0 points and "very severe pain" is graded as 10 points. Pain intensity of "less than 3 points" is indicated as mild pain, "between 3-6 points" as moderate pain, and "more than 6 points" as severe pain. It is seen that the pain increases as the score given increases.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba YILMAZ ESENCAN, Assistant Professor, Study Director — Uskudar University; Sumeyye ÇİFTÇİ, specialist midwife, Principal Investigator — Çam ve Sakura City Hospital
Locations (1):
- Uskudar University Faculty of Health Sciences, Istanbul, Ümraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study will be published in Yöktez.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The work started on May 1 and ended on December 31.
Access Criteria: The study can be accessed by entering Yöktez and typing the name of the study or the names of the administrators.
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/

REFERENCES:
- [Background] Rameshbabu S, Messaoudi SA, Alehaideb ZI, Ali MS, Venktraman A, Alajmi H, Al-Eidi H, Matou-Nasri S. Anastatica hierochuntica (L.) methanolic and aqueous extracts exert antiproliferative effects through the induction of apoptosis in MCF-7 breast cancer cells. Saudi Pharm J. 2020 Aug;28(8):985-993. doi: 10.1016/j.jsps.2020.06.020. Epub 2020 Jul 9. PMID 32792843
- [Background] Ali-Shtayeh MS, Jamous RM, Jamous RM. Plants used during pregnancy, childbirth, postpartum and infant healthcare in Palestine. Complement Ther Clin Pract. 2015 May;21(2):84-93. doi: 10.1016/j.ctcp.2015.03.004. Epub 2015 Apr 2. PMID 25900613
- See also: Fear of Childbirth Scale — https://dergipark.org.tr/tr/download/article-file/752870
- See also: Intervention for Fear of Childbirth: Hypnobirthing — https://gcris.pau.edu.tr/bitstream/11499/6124/1/7ba3f584-23f9-4af0-9a4a-56f72570f94d.pdf
- Available data/document: Individual Participant Data Set: Fear of Childbirth Scale — https://gcris.pau.edu.tr/bitstream/11499/6124/1/7ba3f584-23f9-4af0-9a4a-56f72570f94d.pdf — https://gcris.pau.edu.tr/bitstream/11499/6124/1/7ba3f584-23f9-4af0-9a4a-56f72570f94d.pdf
- Available data/document: Individual Participant Data Set: Fear of Childbirth Scale — https://gcris.pau.edu.tr/bitstream/11499/6124/1/7ba3f584-23f9-4af0-9a4a-56f72570f94d.pdf